CLINICAL TRIAL: NCT06185387
Title: Evaluation of Changes of Renal Morphology, Renal Function and Renal Doppler Parameters Post-percutaneous Nephrolithotomy - A Prospective Case Series Study
Brief Title: Changes Post Percutaneous Nephrolithotomy
Acronym: KUB
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Walid Atef Abdulmonem Abdulhafez, Assistant lecturer, Assiut University
Other Study IDs: Percutaneous*Nephrolithotomy
Record Dates: First submitted 2023-11-12; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Renal Stone
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Using color doppler U/S, Abdominal U/S and radioisotope to evaluate changes of renal morphology, function and doppler parameters post Percutaneous nephrolithotomy

DETAILED DESCRIPTION:
Preoperative assessment:

Detailed history: including history of medical comorbidities, previous history of stone disease or previous treatment of renal stones.

Complete physical examination with measurement and documentation of the pre-operative blood pressure for all patients.

Estimation of body mass index (BMI).

Pre-operative laboratory investigations including:

Complete urine analysis Urine culture and sensitivity test Complete blood picture (CBC). Prothrombin time and prothrombin concentration. Serum urea and creatinine Random blood sugar -Pre-operative imaging investigations: Plain KUB( Number, site, size and radio-opacity of Stones) Abdominal ultrasound ( Dimensions, Shape, borders, contour, orientation & echogenicity, hydronephrosis, stones & others eg. Cysts) Multi-slice computed tomography (MSCT) abdomen and pelvis without contrast. (Dimensions, Shape, borders, contour, orientation, number, site, size, laterality and density of stones) Color Doppler Ultrasonography ( Renal arteries caliber, outline, resistive index, intrarenal arterial waveforms acceleration time& peak systolic velocity) Radioisotope scan (DMSA scan)

-Procedural steps and techniques: Patients with urinary tract infections will be treated with the appropriate antibiotics according to urine culture and sensitivity test until negative culture is obtained.

Percutaneous nephrolithotomy (PCNL) will be performed in prone/supine position under general or spinal anesthesia after insertion of a ureteral catheter to the affected site.

Access will be done under fluoroscopic guidance. Tract dilatation will be done by using either balloon dilator or Amplatz teflon dilators then Amplatz will be inserted.

Stone disintegration after well established track will be done by using either pneumatic or ultrasonic or laser lithotripters.

Stone retrieval will be done by either forceps or Zero-tip dormia basket. At the end of the procedure, plastic tube 22 French may be inserted through the Amplatz sheath as nephrostomy tube or not (tubeless).

Intraoperatively: we record operative time, anaesthesia time, site of renal puncture, puncture relation to last rib, dilatation method, teflon dilatation steps, number of accesses, disintegration methods, use of flexible nephroscope, intraoperative blood transfusion, nephrostomy tube, state of nephrostomy tube when open and perioperative complications.

Post-operative care and follow up:

Plain KUB, abdominal ultrasound, CBC, prothrombin time and concentration & serum creatinine will be done at Day 1 postoperatively.

Measurement of blood pressure at day 1 postoperatively. Abdominal ultrasonography&Color Doppler Ultrasonography at Day 1, Day 7 and Day 90 postoperatively.

Radioisotope scan (DMSA scan) at day 90 postoperatively. Urine analysis

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with age group ≥ 18 years old with renal stones candidate for PCNL.

Exclusion Criteria:

1. Patients with any previous intervention to extract the renal stones.
2. Patients with malrotated/anomalous kidney.
3. Patients with any grade of chronic kidney disease.
4. Patients with bleeding diathesis.
5. Patients who are unfit for surgery.
6. Pregnancy
7. Patients who are refusing the participation in our study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with renal stones that are candidates for PCNL >18 years old
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes of renal function post percutaneous nephrolithotomy | 3 months
  Radioisotope scan (DMSA scan) Split function in %
Changes of renal doppler parameters after percutaneous nephrolithotomy. | 3 months
  Measured by Resistive Index